CLINICAL TRIAL: NCT00133965
Title: Psychosocial Support for Cancer Patients
Status: Completed | Type: Observational
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); University of Manitoba (Other); Edith Cowan University (Other); Visiting Nurse Service of New York (Other)
Responsible Party: William Breitbart, MD, Memorial Sloan Kettering Cancer Center
Other Study IDs: 05-042
Record Dates: First submitted 2005-08-23; First posted 2005-08-24 (Estimated); Last update posted 2011-04-20 (Estimated); Status verified 2011-04

CONDITIONS: Cancer
Keywords: Advanced Cancer; Dignity Care; Supportive Care; Quality of Life; Psychotherapy; Palliative Care
MeSH Terms: conditions — Neoplasms | interventions — Dignity Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (3):
- 1: Dignity Psychotherapy
  Interventions: Behavioral: Dignity Psychotherapy
- 2: Supportive Psychotherapy
  Interventions: Behavioral: Supportive Psychotherapy
- 3: Standard Palliative Care
  Interventions: Behavioral: Standard Palliative Care

INTERVENTIONS:
Behavioral: Dignity Psychotherapy — At the beginning and at the end of the study, you will be asked to fill out a series of questionnaires.will also receive three visits by a mental health professional over a period of five to seven days. You will be asked to fill out some brief questionnaires during this session which ask about feelings about your illness, symptoms, emotional reactions, and support you have available. The second meeting will be scheduled as soon as you are able to do so, within no more than 24 to 48 hours from your initial session with the Research Staff.The third meeting you will also be asked to fill out several questionnaires,including a specific questionnaire regarding your thoughts about the Dignity Psychotherapy Intervention. Total time commitment for this study should be approximately 120-150 minutes.
  Groups: 1
Behavioral: Supportive Psychotherapy — you will receive the standard care you normally would receive, but will also receive three visits by a mental health professional over a period of five to seven days. The initial visit will take approximately 45 minutes. You will be asked to fill out brief questionnaires (described above) during this session.A second contact will be scheduled as soon as you are able to do so, within no more than 24 to 48 hours from your initial session with the research staff. During this second session, you will have the opportunity to discuss with a supportive research therapist issues or topics relevant to your experience of coping with cancer.The third and final contact,you will be asked you to fill out questionnaires similar to those you filled out at the beginning of the study. Total time commitment for this study should be approximately 120-150 minutes.
  Groups: 2
Behavioral: Standard Palliative Care — If you are in the "Standard Palliative Care" group you will receive the standard care that is usually provided here at Memorial Hospital. This can include services such as consultations by physicians, nurses and other healthcare professionals. In addition, referrals to community resources and services can also be made. The study period will be between five and seven days. At the beginning and at the end of the study, you will be asked to fill out a series of questionnaires as described above. Total time commitment for this study should be approximately 60-90 minutes.
  Groups: 3

SUMMARY:
This is an international, 3-site trial (Winnipeg Canada, MSKCC NYC, Perth Australia) accruing 120 patients per site (120x3). The purpose of this study is to compare two types of counseling for cancer patients: "Dignity Psychotherapy" and "Supportive Psychotherapy" as well as "Standard Palliative Care." Many cancer patients seek counseling to help with the emotional burden of their illnesses. Counseling often helps them cope with cancer by giving them a place to express their feelings. We, the investigators at Memorial Sloan-Kettering Cancer Center, have developed a type of counseling we call "Dignity Psychotherapy." It is intended to help cancer patients maintain or enhance a sense of purpose, meaning, and overall quality of life, despite having cancer. "Supportive Psychotherapy" is another type of counseling intended to help patients feel more at ease and express and reflect on any feelings or concerns they might have about their illness. Both of these types of counseling will be compared to "Standard Palliative Care." We will look at how these types of treatments affect patients' mood, outlook, and quality of life. We also want to see how the type of treatment they receive affects their family members and significant others.

DETAILED DESCRIPTION:
Primary Objective:

* To establish the efficacy of a new and unique individual, brief intervention we call "Dignity Psychotherapy" in enhancing a sense of meaning, purpose and overall well-being for patients with advanced, end stage cancer.

Secondary Objectives:

* To compare the effectiveness of "Dignity Psychotherapy" with "Supportive Psychotherapy" and "Standard Palliative Care" in bolstering the patients' sense of meaning, purpose, generativity, and overall sense of dignity and quality of life, while lessening hopelessness, sense of being a burden to others, and suffering.
* To explore the impact "Dignity Psychotherapy" has on the bereavement experience of those family members/significant others taking part in this arm of the study protocol.
* To compare the bereavement experience of bereaved family members/significant others whose loved ones took part in any one of the three study conditions.

ELIGIBILITY:
Inclusion Criteria:

* The patient must be at least 18 years of age (because of the nature of "Dignity Psychotherapy," which presumes a relatively advanced level of social and psychological development).
* Have a terminal illness (Stage IV with a prognosis of less than 6 months, but expected to live at least 7 to 10 days, i.e. the average length of the protocol)
* Must be able to identify a family member/significant other who agrees to participate in the study (in the case of "Dignity Psychotherapy," this family member/significant other will receive the generativity document)
* Be able to communicate with an English-speaking therapist (patients who are visually impaired will be offered assistance with the consent forms and surveys)
* In the investigator's judgement, participant is cognitively able to provide valid, informed consent.

Exclusion Criteria:

* Significant psychiatric disturbance sufficient to preclude participation in a psychotherapeutic intervention (e.g. acute, severe psychiatric symptoms which would require individual treatment and medication management rather than a psychotherapy intervention).
* Active psychotic mental disorder (e.g. schizophrenia, acute mania), or marked paranoid ideation. Patients who are on stable regimens of psychotropic medications (e.g. antidepressants for clinical depression) or who are in concurrent individual or group psychotherapy will not be excluded. This information regarding concurrent psychiatric treatment will be collected and utilized as a co-variate in data analysis.
* Presence of a cognitive disturbance (i.e. delirium or dementia) sufficient to preclude participation in psychotherapy, and/or data collection.
* Physical limitations or illness severity sufficient to preclude participation in psychotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited from the Pain and Palliative Care Service and Gastrointestinal Service of the Memorial Sloan Kettering Cancer Center.
Sampling Method: Non-Probability Sample
Enrollment: 281 (Actual)
Dates: Start 2005-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
To establish the efficacy of a new and unique individual, brief intervention called "Dignity Psychotherapy" in enhancing a sense of meaning, purpose and overall well-being for patients with advanced, end stage cancer | 7-10 days

SECONDARY OUTCOMES:
To compare the effectiveness of "Dignity Psychotherapy" with "Supportive Psychotherapy" and "Standard Palliative Care" in bolstering the patients' sense of meaning | 7-10 days
To explore the impact "Dignity Psychotherapy" has on the bereavement experience of those family members/significant others taking part in this arm of the study protocol | 7-10 days
To compare the bereavement experience of bereaved family members/significant others whose loved ones took part in any one of the three study conditions | Six to nine months following the death of the patient

CONTACTS AND LOCATIONS:
Overall Officials: William Breitbart, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Chochinov HM, Kristjanson LJ, Breitbart W, McClement S, Hack TF, Hassard T, Harlos M. Effect of dignity therapy on distress and end-of-life experience in terminally ill patients: a randomised controlled trial. Lancet Oncol. 2011 Aug;12(8):753-62. doi: 10.1016/S1470-2045(11)70153-X. Epub 2011 Jul 6. PMID 21741309
- See also: Memorial Sloan-Kettering Cancer Center — http://www.mskcc.org